CLINICAL TRIAL: NCT04036916
Title: Sensorimotor Training for Injury Prevention in Collegiate Soccer Players II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: University of West Alabama (Unknown); Mississippi College (Unknown)
Responsible Party: Principal Investigator, Jennifer C. Reneker, Associate Professor, University of Mississippi Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-0157
Record Dates: First submitted 2019-07-23; First posted 2019-07-30 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Concussion, Mild; Sport Injury
Keywords: Concussion; Injury prevention
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality Training (Experimental) (Experimental): Participants will receive multi-modal sensorimotor training interventions, including activities training the vestibular system, oculomotor control and visual perception, neuromotor control and strengthening of the cervical spine, postural control/ balance exercises, and exercises integrating the use of multiple types of sensory information for controlled motor output, including speed and accuracy. Novel headset virtual reality (VR) games/activities; compliant balance surfaces; resistance bands/weight; and biofeedback devices will be utilized to deliver the training intervention. The exercises delivered at each intervention will be delivered in a group format, using a circuit of exercises that each athlete will complete in a session. Subsequent sessions will build upon previous sessions to work the sensorimotor control system in progressively more challenging and sport-specific scenarios. This present study will complete 12 sessions over 6 weeks.
  Interventions: Other: Virtual Reality Sensorimotor Training
- No Virtual Reality Training (Control) (No Intervention): True control.

INTERVENTIONS:
Other: Virtual Reality Sensorimotor Training — Games/activities specifically developed to train the sensorimotor system in headset virtual reality + strengthening of the neck
  Other Names: Cervical strength training
  Arms: Virtual Reality Training (Experimental)

SUMMARY:
The purpose of this project is to evaluate the effectiveness of an injury prevention intervention delivered primarily using headset virtual reality for collegiate soccer players. The hypothesis is that measures of sensorimotor control will improve, injury incidence rate will decrease and on-field soccer performance will improve.

ELIGIBILITY:
Inclusion Criteria:

* Male and female athletes
* 18 years of age or older
* on the soccer roster who are eligible to play in the fall 2019 season at the participating institutions.

Exclusion Criteria:

* Current diagnosis of concussion (i.e. a non-medically cleared concussion)
* Current lower-extremity musculoskeletal injury,
* Seizure disorder with photo sensitivity
* Other medical diagnosis that will prevent participation in the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Injury incidence rate | approximately 16 weeks
  Traumatic injuries (concussion and leg injuries) across the 2019 soccer season/ number of countable athletic exposures
Game Performance | approximately 16 weeks
  Game performance will be analyzed through video recording of the 2019 season's games and analysis of performance metrics (performed by InStat). Key performance indices (with higher scores reflecting better performance during game play) will be used as the metric of game performance.
Standing Balance | Pre to post-intervention (approximately 6 weeks)
  Standing balance (as measured on the Sway balance app 0 - 100 scale)
Reaction Time | Pre to post-intervention (approximately 6 weeks)
  Reaction time (as measured on the Sway balance app) including impulse control; inspection time; and simple reaction time
Oculomotor Control | Pre to post-intervention (approximately 6 weeks)
  Accuracy and latency of saccadic eye movements and smooth pursuit eye movements in response to an object presented to the participant on a computer screen (as measured by the Tobii eye tracker)
Near-Point Convergence | Pre to post-intervention (approximately 6 weeks)
  Distance of point of near-binocular convergence (as measured in centimeters)
Cranial Cervical Flexion Test | Pre to post-intervention (approximately 6 weeks)
  Cranial-cervical flexion neuromotor control (as measured by performance on the Cranial Cervical Flexion Test, mmHg level of control with a 3 second hold on a biofeedback pressure cuff)
Deep Neck Flexor Endurance Test | Pre to post-intervention (approximately 6 weeks)
  Cranial Cervical flexion endurance (measured in seconds)
Isometric Neck Strength | Pre to post-intervention (approximately 6 weeks)
  Measured by a dynamometer in flexion, extension, rotation and side-bending, recorded as force produced in each direction

SECONDARY OUTCOMES:
Score on Smooth Pursuit VR Game | Pre to post-intervention (approximately 6 weeks)
  Score on activities as recorded in headset VR. This game is scored on a 0 - 1000 point scale during completion of the game activity for 60 seconds. Requires participant to follow a moving object with eyes while tracing manually. Accuracy of manual trace produces total score. Higher score = better performance.
Score on Saccades VR Game | Pre to post-intervention (approximately 6 weeks)
  Score on activities as recorded in headset VR. This game is scored on a 0 - 1000 point scale during completion of the game activity for 60 seconds. Requires participant to shift eyes to location of a presented visual stimulus and to activate the location with a manual control. Speed and accuracy of manual activation produces total score. Higher score = better performance.
Score on Near Point Convergence VR Game | Pre to post-intervention (approximately 6 weeks)
  Score on activities as recorded in headset VR. This game is scored on a 0 - 1000 point scale during completion of the game activity for 60 seconds. Requires participant to follow a moving object with eyes while tracing manually. Accuracy of manual trace produces total score. Higher score = better performance.
Score on Joint Position Error VR Game | Pre to post-intervention (approximately 6 weeks)
  Score on activities as recorded in headset VR. This game is scored on a 0 - 1000 point scale during completion of the game activity which is conducted according to the Clinical Joint Position Error Test. Accuracy of head relocation after 3 movements to the left, 3 to the right and 3 into extension produces total score. Higher score = better performance.
Score on Cervical Neuromotor Control VR Game | Pre to post-intervention (approximately 6 weeks)
  Score on activities as recorded in headset VR. This game is scored on a 0 - 1000 point scale during completion of the game activity for 60 seconds. Requires participant to use head and neck movement control to trace a maze. Score is based on accuracy and speed of maze trace.
  Higher score = better performance.
Score on Postural Control (Balance) VR Game | Pre to post-intervention (approximately 6 weeks)
  Score on activities as recorded in headset VR. This game is scored on a 0 - 1000 point scale during completion of the game activity for 60 seconds. Requires participant to maintain standing balance while visual scene in VR is tilting left and right. Score is based on postural sway as recorded by headset sensors. Higher score = better performance.
Score on Cervical Posture VR Game | Pre to post-intervention (approximately 6 weeks)
  Score on activities as recorded in headset VR. This game is scored on a 0 - 1000 point scale during completion of the game activity. Requires participant to reproduce a chin-tucked position and hold for 5 seconds. Score is based on correct head alignment (as compared to starting position, measured by headset sensors) across 10 repetitions. Higher score = better performance.
Score on Visual Figure VR Game | Pre to post-intervention (approximately 6 weeks)
  Score on activities as recorded in headset VR. This game is scored on a 0 - 1000 point scale during completion of the game activity for 60 seconds. Requires participant to visually search a complex scene to find a hidden object. Score is based on the number of correct manual identifications of the hidden object. Higher score = better performance.
Score on Peripheral Vision VR Game | Pre to post-intervention (approximately 6 weeks)
  Score on activities as recorded in headset VR. This game is scored on a 0 - 1000 point scale during completion of the game activity for 60 seconds. Requires participant to focus on central object and use peripheral vision to identify the same object and indicate with a manual selection. Score is based on number of correct identifications. Higher score = better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Reneker, PT, PhD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No
I will have to obtain institutional approval prior to any data being shared externally. This has not been discussed.